CLINICAL TRIAL: NCT00214487
Title: Bifocal Soft Contact Lenses - Do They Slow Progression of Myopia Relative to Single Vision Soft Contact Lenses in Children and Adolescents?
Brief Title: Bifocal Soft Contact Lenses and Their Effect on Myopia Progression in Children and Adolescents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aller, Thomas A., OD (Other)
Collaborators: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas A. Aller, OD, Principal Investigator, Aller, Thomas A., OD
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR-0107
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-06

CONDITIONS: Myopia; Esophoria; Fixation Disparity
Keywords: Myopia Progression; Myopia Control; Bifocal Contact Lenses; Esophoria; Fixation Disparity
MeSH Terms: conditions — Myopia; Esotropia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifocal Contact Lenses (Experimental): Use of bifocal contact lenses to control the progression of myopia
  Interventions: Device: Bifocal Contact Lenses
- Control (Placebo Comparator): Single vision soft contact lenses
  Interventions: Device: Placebo Control

INTERVENTIONS:
Device: Bifocal Contact Lenses — Use of bifocal contact lenses of varying add powers to control the progression of myopia
  Other Names: Bifocal Soft Contact Lenses; Hydrophilic Bifocal Contact Lenses; Simultaneous Vision Bifocal Contact Lenses
  Arms: Bifocal Contact Lenses
Device: Placebo Control — Single vision soft contact lenses
  Other Names: Soft Contact Lenses; Hydrophilic Contact Lenses; Single Vision Soft Contact Lenses
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether bifocal soft contact lenses are effective in controlling the progression of myopia in children and adolescents that exhibit a tendency to excessively cross their eyes while reading (esophoria or eso fixation disparity). Several studies have demonstrated that bifocal or progressive multifocal spectacles are effective in slowing the progression of myopia in children either with near point esophoria and/or with inadequate focusing at near. A prominent theory for one cause of myopia progression is that poorly focused images on the back of the eye (retina) cause the eye to lengthen, causing an increase in myopia. Bifocal contact lenses may reduce this retinal defocus, reducing the stimulus to eye elongation, and thus may reduce myopia progression.

DETAILED DESCRIPTION:
Myopia has become the focus of growing attention and concern because the prevalence of myopia appears to increasing in some populations (reaching 90% for some university student populations in Asia). There are serious risks to higher levels of myopia, including cataracts, glaucoma, retinal detachment and myopic retinal degeneration. Several studies have shown mild to moderate control of myopia progressionwith bifocal or multifocal spectacles in children with esophoria at near and/or with accommodative deficiencies. Pilot studies by the P.I. have suggested that bifocal contact lenses may control myopia progression in children with near point eso fixation disparity.

CONTROL is a controlled, randomized, prospective, double-blind, one year study of the changes in myopia in 80-90 subjects from age 8-18 with low to moderate levels of myopia, low levels of astigmatism, and eso fixation disparity at near, when fitted with either bifocal soft contact lenses or single vision soft contact lenses. The primary outcome measures will be cycloplegic refraction and axial length measures.

ELIGIBILITY:
Inclusion Criteria:

* Myopia between -0.50 and -6.00
* Eso fixation disparity at 33cm with distance correction
* Astigmatism 1.00 or less
* Ability to wear soft contact lenses

Exclusion Criteria:

* Presence of ocular disease preventing wear of contacts
* Pregnancy or nursing
* Use of certain medications

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2003-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A. Aller, O.D., Principal Investigator

REFERENCES:
- [Background] Aller TA, Wildsoet C. Bifocal soft contact lenses as a possible myopia control treatment: a case report involving identical twins. Clin Exp Optom. 2008 Jul;91(4):394-9. doi: 10.1111/j.1444-0938.2007.00230.x. PMID 18601670
- [Background] Tarrant J, Severson H, Wildsoet CF. Accommodation in emmetropic and myopic young adults wearing bifocal soft contact lenses. Ophthalmic Physiol Opt. 2008 Jan;28(1):62-72. doi: 10.1111/j.1475-1313.2007.00529.x. PMID 18201337
- [Background] Aller TA. Design of a prospective clinical trial of the use of bifocal soft contact lenses to control myopia progression (CONTROL). Proceedings of the 10th International Myopia Conference 2004:29.
- [Result] Aller TA, Wildsoet C. Results of a one-year prospective clinical trial (CONTROL) of the use of bifocal soft contact lenses to control myopia progression. Ophthalmic and Physiological Optics 26(S1), 8-9.
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645
- See also: Click here for more information about the CONTROL Study — http://www.draller.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bifocal Contact Lenses | Control
Started | 43 | 43
Completed | 38 | 40
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Population: Numbers reflect those subjects screened, enrolled, randomized with at least one follow up examination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bifocal Contact Lenses | Control | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 38 | 40 | 78
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Changes in Cycloplegic Autorefraction in One Year.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Bifocal Contact Lenses | Control
Number analyzed (Participants) | 38 | 40
Diopters | -0.22 (0.34) | -0.78 (0.45)

2. Secondary Outcome: Keratometric Changes at One Year.
Time Frame: One year
Reporting Status: Not Posted

3. Secondary Outcome: Changes in Manifest Refraction at One Year.
Time Frame: One year
Reporting Status: Not Posted

4. Secondary Outcome: Relationship Between Residual Fixation Disparity and Myopia Progression.
Time Frame: One year
Reporting Status: Not Posted

5. Secondary Outcome: Changes in Cycloplegic Subjective Refraction in One Year
Time Frame: One year
Reporting Status: Not Posted

6. Secondary Outcome: Changes in Axial Length at One Year.
Time Frame: One year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Bifocal Contact Lenses | Control
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator acknowledges that the data to be collected is proprietary. The Investigator agrees not to publish, divulge, reveal, disclose or otherwise make available, the data to others without the permission of sponsor unless the data have already been, or are subsequently published or disclosed by order of a court of law. The Investigator will not be free to publish papers dealing with the results of any Research performed under this Agreement without the consent of sponsor.